CLINICAL TRIAL: NCT07084038
Title: Effect of Glycosuria on Urinary Protein in Patients With Chronic Kidney Disease Treated With SGLT2 Inhibitor
Brief Title: Effect of Glycosuria on Urinary Protein in Patients With Chronic Kidney Disease Treated With SGLT2 Inhibitors
Status: Active, not recruiting | Type: Observational
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, Principal Investigator, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2025-295-01
Record Dates: First submitted 2025-07-22; First posted 2025-07-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial aims to investigate the correlation between glycosuria levels and urinary protein in chronic kidney disease patients treated with Sodium-Glucose Transporter 2 Inhibitors(SGLT2i), and to explore whether glycosuria can reflect the therapeutic response to SGLT2i in these patients. Through this study, the investigators hope to provide some clinical references for optimizing SGLT2i dosing strategies.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years. Patients with a confirmed diagnosis of chronic kidney disease (CKD). Currently receiving stable, standard-dose SGLT2i therapy at screening. Proteinuria ≥0.15 g/24 h (or urine protein-to-creatinine ratio [UPCR] ≥440 mg/g or urine albumin-to-creatinine ratio [UACR] ≥300 mg/g) at screening.

Estimated glomerular filtration rate (eGFR) ≥15 mL/min/1.73m² calculated by the CKD-EPI creatinine equation at screening.

Willing and able to provide written informed consent.

Exclusion Criteria:

Discontinuation of SGLT2i during the follow-up period. History of symptomatic hypotension (systolic blood pressure<90 mmHg) without antihypertensive medication, or current hypotensive episode at screening.

Unstable renal function (e.g., acute kidney injury or rapidly progressive glomerulonephritis with a >50% decline in eGFR within 3 months prior to screening).

Use of corticosteroids or having an indication for corticosteroid therapy within the past 6 months.

Receipt of immunosuppressive therapy or having an indication for immunosuppressive therapy within the past 6 months.

History of intolerance to SGLT2 inhibitors. History of ketoacidosis within the past 5 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years diagnosed with chronic kidney disease (CKD) at the First Medical Center of the PLA General Hospital by March 2026, who regularly received oral administration of standard-dose SGLT2 inhibitors (SGLT2i), will be included. Medical records and laboratory test results (including routine blood tests and blood biochemical parameters) will be collected. Changes in 24-hour urinary glucose and urinary protein levels from baseline will be observed at 3 and 6 months after SGLT2i administration.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change in urinary protein from baseline at 3 months and 6 months of follow-up | 3 months and 6 months
  The percentage change in urinary protein from baseline at 3 months and 6 months of follow-up

SECONDARY OUTCOMES:
The proportion of a 50% reduction in urinary protein, the proportion of a 30% reduction in urinary protein, and the changes in estimated glomerular filtration rate (eGFR) | 3 months and 6 months
  The proportion of patients with a 50% reduction in urinary protein and a 30% reduction in urinary protein at 3 months and 6 months of follow-up, as well as the percentage change in estimated glomerular filtration rate (eGFR).

CONTACTS AND LOCATIONS:
Overall Officials: Guangyan Cai, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital,, Beijing, Beijing Municipality, China